CLINICAL TRIAL: NCT03359694
Title: Mutation Scores and Differential Protein Evaluating Efficacy in Neo-adjuvant Chemotherapy and the Non-PCR Patients Treated With Sequential Nalvelbine and Xeloda in HER2(-) Luminal B Breast Cancer
Brief Title: Mutation Scores and Differential Protein Evaluating Efficacy in Adjuvant Chemotherapy in HER2(-) Luminal B Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NO20170819
Record Dates: First submitted 2017-11-20; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Susceptibility, Genetic; Chemotherapy Effect
Keywords: breast cancer, neoadjuvant chemotherapy,susceptible gene
MeSH Terms: conditions — Genetic Predisposition to Disease; Breast Neoplasms | interventions — liposomal doxorubicin; Docetaxel; Vinorelbine; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- DT group (Experimental): Pegylated liposomal doxorubicin and Docetaxel Treatment group Pegylated liposomal doxorubicin 30mg/m2，iv，d1， Docetaxel 75mg/m2，iv，d1， q21d×6
  Interventions: Drug: DT group
- ET group (Active Comparator): Conventional doxorubicin and Docetaxel Treatment group Conventional doxorubicin 75mg/m2，iv，d1， Docetaxel 75mg/m2，iv，d1， q21d×6
  Interventions: Drug: ET group
- NX group (Experimental): Navelbine and Xeloda treatment group in group of Non-pCR patients Navelbine IVD 25 mg/m2 D1、D8 Xeloda PO 1000 mg/m2 bid D1-D14 q21d×4
  Interventions: Drug: NX group
- Control group (No Intervention): no treatment group of Non-pCR patients after DT or ET neoadjuvant chemotherapy.
  No drugs treatment in this group.

INTERVENTIONS:
Drug: DT group — Pegylated liposomal doxorubicin 30mg/m2，iv，d1， Docetaxel 75mg/m2，iv，d1， q21d×6
  Other Names: Pegylated liposomal doxorubicin and Docetaxel
  Arms: DT group
Drug: ET group — Conventional doxorubicin 75mg/m2，iv，d1， Docetaxel 75mg/m2，iv，d1， q21d×6
  Other Names: Conventional doxorubicin and Docetaxel
  Arms: ET group
Drug: NX group — Navelbine IVD 25 mg/m2 D1、D8 Xeloda PO 1000 mg/m2 bid D1-D14 q21d
  Other Names: Navelbine and Xeloda
  Arms: NX group

SUMMARY:
We plan to carry out a prospective, randomized, open phase III clinical trial which sponsored by the Tianjin Medical University Cancer Hospital and Institute. The primary aim is to evaluate pCR of DT and ET regimen as neoadjuvant chemotherapy in the treatment of HER2 negative Luminal B breast cancers and the correlation of pCR respectively with the susceptible gene mutation scores and differential protein identified by proteomics. For patients with pCR, the association between the 5 year DFS and susceptible gene mutation scores and differential protein identified by proteomics will be evaluated. All Non-pCR patients will receive NX chemotherapy for 4 cycles, and to evaluate correlations between 5 year DFS of these patients respectively with susceptible gene mutation scores and differential protein identified by proteomics, and to evaluate the safety of neoadjuvant chemotherapy and sequential adjuvant NX regimen therapy. Meanwhile, we will verify susceptible gene mutation scores and differential protein identified by proteomics are significant predictors of HER2 negative Luminal B breast cancer chemotherapy sensitivity and prognosis, and explore the feasibility of susceptible gene mutation scores and differential protein in clinical application.

DETAILED DESCRIPTION:
This is a prospective, randomized, open phase III clinical trial which will be sponsored by the Tianjin Medical University Cancer Hospital and Institute. The primary aim is to evaluate pCR of Pegylated Liposomal Doxorubicin and Docetaxel (DT) Compared to Conventional Doxorubicin and Docetaxel (ET) regimen as neoadjuvant chemotherapy in the treatment of HER2 negative Luminal B breast cancers and the correlation of pCR respectively with the susceptible gene mutation scores and differential protein identified by proteomics. For patients with pCR, the association between the 5 year DFS and susceptible gene mutation scores and differential protein identified by proteomics will be evaluated. All Non-pCR patients will receive NX chemotherapy for 4 cycles, and to evaluate correlations between 5 year DFS of these patients respectively with susceptible gene mutation scores and differential protein identified by proteomics, and to evaluate the safety of neoadjuvant chemotherapy and sequential adjuvant Nalvelbine and Xeloda (NX) regimen therapy. Meanwhile, we will verify susceptible gene mutation scores and differential protein identified by proteomics are significant predictors of HER2 negative Luminal B breast cancer chemotherapy sensitivity and prognosis, and explore the feasibility of susceptible gene mutation scores and differential protein in clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Compliance with test procedures and good compliance
* Females, Age more than 18 years of age, less than 70 years old
* The ECOG score is 0-1
* Primary invasive cancer, T2-4bN0-2M0 breast cancers
* Neoadjuvant chemotherapy with standard 6 courses should be completed
* Patients must undergo standard breast cancer surgery after neoadjuvant chemotherapy
* Luminal B, Her2 negative patients
* No other malignant tumors occurred at the same time
* adequate liver and kidney function

Exclusion Criteria:

* Any metastasis
* Suffered other maligant tumors
* Participate in other trials
* Accompanied with severe systemic disease and / or uncontrollable infection
* Pregnant and lactating women
* Dysfunction of liver and kidney

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 2 years
  pCR rate in the DT and ET group

SECONDARY OUTCOMES:
Efficacy of neo-adjuvant chemotherapy | 5 years
  5-year DFS in the DT and ET group
Efficacy of sequential chemotherapy | 6 years
  5-year DFS of non- pCR patients treated by sequential NX regimen

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhang, Doctor, Principal Investigator — Tianjin Medical University Cancer Institure and Hospital
Locations (1):
- Jin Zhang, Tianjin, China

IPD SHARING:
Plan to Share IPD: No